CLINICAL TRIAL: NCT03495128
Title: Determination of the Time-course of Development of Insulin Resistance, and Associated Molecular and Muscular Adaptations, During Inactivity in 3 Days of Bed-rest
Brief Title: Metabolic and Muscular Adaptations During Inactivity in 3 Days of Bed-rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6-1704; BB/P005004/1 (Other Grant/Funding Number: BBSRC)
Record Dates: First submitted 2018-03-30; First posted 2018-04-11 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Muscle Atrophy; Insulin Sensitivity
Keywords: muscle protein breakdown; inactivity; bed rest
MeSH Terms: conditions — Muscular Atrophy; Insulin Resistance; Sedentary Behavior | interventions — Bed Rest

STUDY DESIGN:
Intervention Model Description: longitudinal assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bed rest (Experimental): Three days of bed rest at -6 degrees of head-down tilt
  Interventions: Other: Bed Rest
- Reconditioning (Experimental): Three days of one-legged knee extension contractions to recondition one leg
  Interventions: Other: Reconditioning

INTERVENTIONS:
Other: Bed Rest — 3 days of head down tilt (-6 degrees) bed rest
  Arms: Bed rest
Other: Reconditioning — daily resistance training (for 3 days) on one leg
  Arms: Reconditioning

SUMMARY:
Space flight is associated with detrimental changes to the human body, including bone and muscle loss, fluid changes and deconditioning of muscles in the heart and blood vessels. Bed rest experiments, on Earth, are used to study these changes in healthy volunteers, as the disuse of muscles, and impact on the body, mimic the changes seen in the low-gravity environment of Space. Moreover, these changes are similar to those reported in people who remain in bed for long periods of time, such as is seen in intensive care or stroke patients, and bed rest studies also allow the physiological and biochemical impacts of this confinement to be investigated. For example, we know from previous research that muscle inactivity can lead to the development of resistance to the action of the hormone 'insulin', which is a longer term risk factor for the development of type 2 diabetes. Previous studies suggest that this inactivity-induced insulin resistance occurs within the first 48 hours of immobilization. However, it is not clear whether the biochemical and physiological processes underlying these short-term responses to inactivity are the same as those seen in the longer term. The current study aims to investigate the biochemical and physiological changes seen after 3 days of bed rest and to compare to those measured in a previous 57 days bed rest study carried out at Institut Médecine Physiologie Spatiale (MEDES; Toulouse, France). A 3-day period of reconditioning will subsequently be used to determine if these changes can be readily reversed.

DETAILED DESCRIPTION:
Bed rest is a widely accepted experimental model used to study physiological adaptations to space flight, including bone and muscle mass loss, fluid shift, and cardiovascular deconditioning. Generally, participants are asked to spend a period in bed, with all activities of daily living being performed in a horizontal or head-down tilt (HDT) position, thus minimising use of all muscles and bringing about significant physiological adaptations similar to those observed during space flight. A substantial number of human bed rest studies have been performed ranging from 3-370 days duration. However, there are currently gaps in our understanding of; the rate and magnitude of the physiological dysregulation that occurs during actual and simulated microgravity (as most studies to date have considered mainly pre and post-bed rest time-points); the sites and mechanisms controlling bed rest-induced dysregulation; whether the processes underlying acute physiological changes are the same as those seen in the longer term. Improving our understanding of these issues would enable interventions aimed at minimizing bed-rest induced physiological dysregulation to be most effectively focused on time periods when the rate of onset of physiological dysregulation is likely to be at its greatest. This would then contribute to future success being achieved in prolonged human space flight, e.g. a manned mission to Mars, because an understanding of the aetiology and time-course of the physiological dysregulation that accompanies prolonged exposure to microgravity would enable effective counter-measures to be implemented. Furthermore, bed rest models present a unique opportunity to study the consequences of bed rest on those who may sustain prolonged periods of inactivity during hospitalisation, arising from illness or injury.

Inactivity is associated with the development of insulin resistance and contributes to the development of many modern metabolic diseases including obesity, type 2 diabetes, dyslipidaemia and hypertension (1,2); with physical inactivity being cited as the principal cause of 27% of diabetes and 30% of ischaemic heart disease cases. However, the time course, relative tissue specificity (liver vs muscle) and mechanistic basis of inactivity induced insulin resistance, and its reversal by remobilisation, represent major gaps in our current understanding. Furthermore, insulin resistance is an observation with several possible aetiologies and the mechanisms involved in the development of this condition with short term bedrest/immobilisation may be different to those involved with longer term / chronic inactivity. Further research in this area is therefore warranted.

The current study is part of a larger project which includes a 60 day, long term, bed rest study conducted in collaboration with the European Space Agency, at the Institut Médecine Physiologie Spatiale facility in Toulouse, France, and will be compared to the measures being conducted in the long term bed rest experiment.

'Run-in' phase; Following a successful medical screening, participants will start a 'Run-in' phase during which their habitual activity levels will be assessed by accelerometry. Individualised energy requirements will be estimated using the modified Harris-Benedict resting metabolic rate equation and physical activity level factor and a standardised diet (macronutrient composition (expressed as a percentage of total dietary energy intake) being ~55% carbohydrates, ~30% fat and ~15% protein) will be provided for the 3-days preceding the first experimental session. The day before this session, participants will be asked to abstain from any strenuous exercise and to fast from midnight, consuming only water from that time. On arrival, a dual-energy X-ray absorptiometry (DEXA) scan will be carried out to characterise whole body and leg fat masses. The participant will then be asked to lie on a hospital bed in the supine position (one pillow) and muscle volume and architecture measurements will be determined by ultrasound imaging of the vastus lateralis muscle using a 100 mm linear array 13-4 megahertz probe. This will provide a global representation of quadriceps muscle anatomy in order to standardise calculations of leg glucose uptake and determine the contribution of muscle mass and intramyocellular lipid to leg insulin resistance. Muscle biopsy samples will be obtained from the vastus lateralis before and immediately after a 3hr hyperinsulinemic euglycemic clamp (3). Muscle biopsies will be obtained using the Bergström technique under sterile conditions, after injection of local anaesthetic. An anterograde femoral venous catheter will be inserted (using the Seldinger technique under ultrasound guidance) to enable venous blood draining from the leg to be analysed for glucose concentration and compared with the glucose concentration of arterialised-venous blood samples (Time points 0, 150, 160, 170 and 180 mins). At the same time as the femoral venous blood sample is taken, a femoral artery blood flow assessment (mmol/min) will be made using ultrasonography to enable leg glucose uptake to be calculated. Indirect calorimetry will be performed before and in the last 15 minutes of the 180min hyperinsulinaemic-euglycaemic clamp.

The day after the 'clamp' visit, a 3 Tesla magnetic resonance spectroscopy (MRS) scan will be undertaken to assess intramyocellular lipid (IMCL), extramyocellular lipid (EMCL), and hepatic triglyceride content. A magnetic resonance imaging (MRI) scan will also be performed to determine mid-thigh muscle cross-sectional area and whole body muscle mass. Following the magnetic resonance (MR) scans, participants will undergo a short lower limb proprioceptive assessment on a specially designed somatosensory apparatus called the Active Movement Extent Discrimination Assessment (AMEDA). Participants will stand on the apparatus and have each ankle moved through 5 different angles of inversion and are asked to rate the degree of ankle position. This method has been validated to determine proprioceptive discrimination and will be repeated after the MR performed on day 4 to assess differences before and after bed rest.

Before the bed rest period begins, saliva and urine samples will be collected for measures of background labelling of creatine, creatinine, water and 3-methylhistidine (MH) with deuterium. Following this, participants will be provided with a drink containing stable isotope tracers; deuterated creatine (D3-Creatine 30 mg; to measure whole body muscle mass) and deuterated, or 'heavy', water (D2O, 3g/kg body weight, divided into 3 aliquots ingested 20 min apart, to measure muscle protein synthesis (MPS) from muscle tissue incorporation measurements). Two hours after consumption of the final D2O dose, a saliva sample will be collected to measure the equilibration of D2O throughout the body water pool. A 24h urine collection will be carried out in the 24hrs post D3-creatine ingestion, and a spot urine sample will be taken at 36hr, 48hr and 72h. Urine will be analysed for D3-creatine to account for 'spillover', and D3-creatinine labelling which will reflect dilution of label in the whole body creatine pool. Total body creatine pool size and muscle mass will be calculated from the D3-creatinine enrichment in urine at 72h, after accounting for any loss of D3 creatine straight into urine. In addition, 24 hours prior to starting bed rest (day -1), participants will ingest Methyl-D3-3 methylhistidine (10mg, D3-MH to measure whole body muscle myofibrillar breakdown) tracer in a drink. A further 10mg will be given on day 2 of bed rest, with blood monitoring on day 3.

Bed rest Phase; Participants will arrive at the facility at 8am on the morning of day 1 following an overnight fast from 22:00 the evening before. For simulation of the physiological effects of microgravity, the bed is maintained in a 6° head down tilt position (HDT- position). A Bard microneedle muscle biopsy will be performed and repeated on the following morning (day 2 of bed rest) to assess cumulative muscle protein synthesis over the first 24 hours of bed rest. On each day following the biopsy, an anterograde venous cannula will be inserted into the arm for sampling of blood every hour for a total of 6 hours for the measurement of D3-MH labelling.

Top-ups of D2O (calculated from water turnover rates) will be provided to participants on days 1 and 3 of bed rest, to maintain D2O enrichment. A saliva sample will be taken to measure D2O body water enrichment and a urine sample for D3 Creatinine labelling.

During bed rest, participants will remain in bed for 24h a day. All activities of daily living such as hygienic procedures, eating, reading and 'going' to the bathroom (use of bed-pans and urine bottles) take place whilst maintaining the head down position for the duration of the study. Participants are allowed to move from side to side (from supine to ventral or lateral positions), but are not allowed to sit up or stand at any time. The use of one small size flat pillow is allowed as long as the shoulders still touch the mattress. Dietary intake will be controlled, with an activity multiplier of 1.2 being used to determine daily energy intake requirements. Five daily meals (breakfast, morning snack, lunch, afternoon snack and dinner) are served at the same time of the day, throughout. The participants are encouraged to consume all the food provided. They can consume less than provided, but will not receive any additional food. Each food item is weighed on a precision (±0.1 g) scale and where participants do not eat all food given, the unconsumed food items is re-weighed and the value subtracted from the initial weight to provide actual food intake. Subjects keep a strict day-night cycle. They are woken at 7:00 am and lights out occurs at 11:00pm.

On the morning of day 4, after an overnight fast, the participants will undergo the second 'clamp' day as described above (ultrasound scan of the thigh, indirect calorimetry, femoral vein cannulation, muscle biopsies and an euglycemic hyperinsulinemic clamp). After this, gradual, supervised return to 'upright' in the bed will be carried out, with continuous cardiovascular monitoring to avoid postural hypotension. Participants will remain in bed but will be allowed to sit in the upright position until the morning of day 5.

Post bed-rest phase; The morning of day 5, participants will transfer (without weight-bearing) into a wheelchair, then transported to the 3 Tesla MR scanner for their post bed rest MR scans. They will be required to be fasted from 22:00 the evening before. Following the MR scans, participants will be fed and allowed to return to standing in a controlled environment. They will then undergo supervised rehabilitation in the University of Nottingham gym facilities comprising of 6 sets of 8 repetitions (at 75% of maximum) of one-legged knee extension contractions on a randomly allocated leg, as this has been shown to provide an anabolic stimulus (4), and then be allowed to return home. Rehabilitation sessions will last approximately 30 minutes. They will return on days 6 and 7 of the non-bed rest period to undergo further supervised rehabilitation sessions as above. Standardised dietary intake will be maintained throughout the post bed rest phase. At 08:00 on the morning of day 8 they will attend the laboratory to undergo a final 'clamp' visit consisting of the same procedures detailed above, with the following modification; a Bergström muscle biopsy will be performed on the leg that underwent rehabilitation exercise training pre and post euglycemic hyperinsulinemic clamp. A Bard microneedle biopsy will be performed on the contralateral leg only before the 3hr clamp, in order to compare muscle protein synthesis between legs. Finally, on day 9 the MRS and MRI scans will be performed in the same manner described above. When the final MRS scan has been performed that will be the end of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy participants
* Body mass index 20 - 26 kg/m2
* Height 158 - 190 cm (62 - 75 inches),
* Participants that are able to consent to participation in the entire study
* Signed informed consent

Exclusion Criteria:

* regular use of prescribed or 'over-the counter' medication
* Bone mineral density (measured by Dual-Energy X-ray Absorptiometry) more than 1.5 standard deviation less than t-score
* Family history of thrombosis or positive response in thrombosis blood screening: Antithrombin III, High sensitive C-Reactive Protein, protein kinase B, F-V-Leiden, Prothrombin mutation, Lupus-prothrombin time, Factor II
* Any current medical condition
* A medical history of thyroid dysfunction, renal function disorder (including renal stones), diabetes, cardiac arrhythmias and cardiovascular disorders, migraines, allergies, hypertension, hypocalcaemia, uric acidaemia, lipidemia or hyperhomocysteinemia, hiatus hernia, bowel surgery or gastro-oesophageal reflux
* History of a mental health disorder
* Smoker within six months prior to the start of the study
* Dependence on drugs, medicine or alcohol
* History of orthostatic intolerance, vestibular disorders or claustrophobia
* Special food diet, vegetarian or vegan, history of intolerance to lactose or food allergy,
* Osteosynthesis material, presence of metallic implants, history of knee problems or joint surgery/broken leg,
* Orthopaedic or musculoskeletal disorders.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Insulin stimulated whole body glucose uptake | after 3 days of bed rest, compared to pre-bed rest
  Determined during a hyperinsulinemic, euglycemic clamp

SECONDARY OUTCOMES:
Change in Insulin stimulated whole body glucose uptake | after 3 days of reconditioning, compared to post-bed rest
  Determined during a hyperinsulinemic, euglycemic clamp
Change in Insulin stimulated leg glucose uptake | after 3 days of bed rest, compared to pre-bed rest
  Determined during a hyperinsulinemic, euglycemic clamp, using arterialised-venous vs. venous difference in glucose concentration and ultrasound derived femoral artery blood flow
Change in Insulin stimulated leg glucose uptake | after 3 days of reconditioning, compared to post- bedrest
  Determined during a hyperinsulinemic, euglycemic clamp, using arterialised-venous vs. venous difference in glucose concentration and ultrasound derived femoral artery blood flow
Change in Whole body muscle mass | after 3 days of bed rest, compared to pre-bed rest
  Determined using whole body magnetic resonance imaging
Change in Whole body muscle mass | after 3 days of reconditioning, compared to post- bed rest
  Determined using whole body magnetic resonance imaging
Change in Muscle Pyruvate dehydrogenase activity | after 3 days of bed rest, compared to pre-bed rest
  Determined biochemically from vastus lateralis muscle biopsy samples before (fasting state) and at the end of the 3hr hyperinsulinemic, euglycemic clamp (insulin stimulated state).
Change in Muscle Pyruvate dehydrogenase activity | after 3 days of reconditioning, compared to post- bed rest
  Determined biochemically from vastus lateralis muscle biopsy samples before (fasting state) and at the end of the 3hr hyperinsulinemic, euglycemic clamp (insulin stimulated state).
Change in Muscle gene expression | after 3 days of bed rest, compared to pre-bed rest
  expression of genes related to protein turnover, fuel metabolism, in muscle biopsy samples from vastus lateralis taken before (fasting state) and at the end of the 3hr hyperinsulinemic, euglycemic clamp (insulin stimulated state)
Change in Muscle gene expression | after 3 days of reconditioning, compared to post-bed rest
  expression of genes related to protein turnover, fuel metabolism, in muscle biopsy samples from vastus lateralis taken before (fasting state) and at the end of the 3hr hyperinsulinemic, euglycemic clamp (insulin stimulated state)
Change in Muscle protein turnover | after 3 days of bed rest, compared to pre- bedrest
  oral administration of stable isotopes Methyl-D3-3 methylhistidine, D3 creatine and D2O will be used to assess muscle protein breakdown and muscle protein synthesis (urine, saliva, blood and muscle biopsy analysis)
Change in muscle triglyceride content | after 3 days of bed rest, compared to pre-bed rest
  Determined using mid-thigh magnetic resonance spectroscopy
Change in muscle triglyceride content | after 3 days of reconditioning, compared to post-bed rest
  Determined using mid-thigh magnetic resonance spectroscopy
Change in liver triglyceride content | after 3 days of bed rest, compared to pre-bed rest
  Determined using magnetic resonance spectroscopy of the liver
Change in liver triglyceride content | after 3 days of reconditioning, compared to post-bed rest
  Determined using magnetic resonance spectroscopy of the liver
Change in Markers of bone turnover | after 3 days of bed rest, compared to pre-bed rest
  biochemical analysis of blood and urine; procollagen I protein, Calcium, Albumin, ionized calcium, Parathyroid hormone, Dickkopf-1, Sclerostin, carboxy-terminal collagen crosslinks, Osteocalcin
Change in Markers of bone turnover | after 3 days of reconditioning, compared to post-bed rest
  biochemical analysis of blood and urine; procollagen I protein, Calcium, Albumin, ionized calcium, Parathyroid hormone, Dickkopf-1, Sclerostin, carboxy-terminal collagen crosslinks, Osteocalcin
change in adipose tissue function | after 3 days of bed rest, compared to pre-bed rest
  biochemical analysis of blood; Adiponectin, Leptin, Visfatin, Resistin
change in adipose tissue function | after 3 days of reconditioning, compared to post-bed rest
  biochemical analysis of blood; Adiponectin, Leptin, Visfatin, Resistin

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Greenhaff, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Laboratories, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergouignan A, Rudwill F, Simon C, Blanc S. Physical inactivity as the culprit of metabolic inflexibility: evidence from bed-rest studies. J Appl Physiol (1985). 2011 Oct;111(4):1201-10. doi: 10.1152/japplphysiol.00698.2011. Epub 2011 Aug 11. PMID 21836047
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Brook MS, Wilkinson DJ, Mitchell WK, Lund JN, Phillips BE, Szewczyk NJ, Greenhaff PL, Smith K, Atherton PJ. Synchronous deficits in cumulative muscle protein synthesis and ribosomal biogenesis underlie age-related anabolic resistance to exercise in humans. J Physiol. 2016 Dec 15;594(24):7399-7417. doi: 10.1113/JP272857. Epub 2016 Nov 7. PMID 27654940
- [Result] Shur NF, Simpson EJ, Crossland H, Chivaka PK, Constantin D, Cordon SM, Constantin-Teodosiu D, Stephens FB, Lobo DN, Szewczyk N, Narici M, Prats C, Macdonald IA, Greenhaff PL. Human adaptation to immobilization: Novel insights of impacts on glucose disposal and fuel utilization. J Cachexia Sarcopenia Muscle. 2022 Dec;13(6):2999-3013. doi: 10.1002/jcsm.13075. Epub 2022 Sep 4. PMID 36058634